CLINICAL TRIAL: NCT07356973
Title: Open-label Phase 2 Safety and Efficacy Trial of Irinotecan-ChemoSeed Administered Directly Into the Resection Margin in Patients With Surgically Resectable Glioblastoma
Brief Title: Irinotecan-ChemoSeed in Surgically Resectable Glioblastoma
Acronym: OPTICAL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CRISM Therapeutics LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICS1; IRAS ID: 1012556 (Registry Identifier: Regulatory Agency Identifier)
Record Dates: First submitted 2026-01-13; First posted 2026-01-21 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Determination (Part 1) (Other): Dose escalation to identify maximum tolerance dose MTD
  Interventions: Drug: irinotecan-ChemoSeed implementation into the resection cavity after surgical resection of GBM
- Efficacy Testing (Part 2) (Other): 2 : 1 randomization irinotecan-ChemoSeed versus standard of care
  Interventions: Drug: irinotecan-ChemoSeed implementation into the resection cavity after surgical resection of GBM

INTERVENTIONS:
Drug: irinotecan-ChemoSeed implementation into the resection cavity after surgical resection of GBM — irinotecan-ChemoSeed implementation into the resection cavity after surgical resection of GBM

SUMMARY:
Part 1 (dose escalation, safety, and preliminary efficacy) Part 1 is a non-randomised, single-arm design in 12 participants with recurrent GBM suitable for maximal safe surgical resection.

Part 1 will evaluate safety, determine the MTD of irinotecan-ChemoSeed and the RP2D (corresponding to coverage of as much of the resection cavity as possible, up to the MTD) and evaluate efficacy. All Part 1 participants will be administered irinotecan- ChemoSeed concurrent to Standard of Care (SoC) treatment. Part 1 dose- escalation will start at 72 mg of IRN Part 2, in 135 participants with newly diagnosed GBM suitable for maximal safe surgical resection, will assess the efficacy of irinotecan-ChemoSeed. The actual number of irinotecan-ChemoSeeds administered into the resected tumour margin of the tumour cavity after surgical resection will be at the discretion of the neurosurgical consultant up to the MTD, to cover as much of the resection cavity as possible. Participants will be randomised in a 2:1 ratio:

* Arm 1: Irinotecan-ChemoSeed +SoC: Irinotecan-Chemoseeds administered into the resection margin following maximal safe surgical resection, with fractionated RT, concomitant and maintenance TMZ (based on Stupp protocol) starting 4 to 6 weeks after surgery per institution standard practice.
* Arm 2: SoC treatment only: maximal safe surgical resection with fractionated RT, concomitant and maintenance TMZ (based on Stupp protocol) starting 4 to 6 weeks after surgery per institution standard practice.

ELIGIBILITY:
Inclusion Criteria:

* 1. Radiologically relapsed, neuropathologically verified GBM (by the WHO 2021 criteria) (Part 1) or newly diagnosed, radiologically suspected GBM (Part 2) amenable to surgical resection.

  2. Male or female aged 18 years or older. 3. Ability to understand and the willingness to sign a written informed consent form (ICF).

  4. KPS ≥ 70. 5. Life expectancy ≥ 6 months. 6. Adequate organ and marrow function as follows (all required):
  1. Absolute neutrophil count ≥ 1.5 k/µL
  2. Platelets ≥ 100 k/µL
  3. Haemoglobin ≥ 9 g/dL
  4. Serum creatinine ≤ 1.8 mg/dL or creatinine clearance > 50 mL/min
  5. Bilirubin ≤ 1.5 mg/dL
  6. Alanine aminotransferase (ALT) ≤ 3.0 × upper limit of normal (ULN)
  7. Aspartate aminotransferase (AST) ≤ 3.0 × ULN
  8. Prothrombin time ≤ 1.5 × ULN
  9. International normalised ratio (INR) ≤ 1.5 × ULN
  10. Partial thromboplastin time ≤ 1.5 × ULN 7. Women of childbearing potential must agree to use a highly effective method of contraception for the duration of the trial or for 5X the systemic half-life (i.e., 6 weeks) plus 6 months following irinotecan-ChemoSeed administration, whichever is the longest.. Female participants must refrain from egg donation during the same time period. 8. Male participants of reproductive potential, who intend to be sexually active with a female partner of childbearing potential, must commit to use barrier contraception (e.g., condom) for the duration of the trial or for 5X the systemic half-life (i.e., 6 weeks) plus 6 months following irinotecan-ChemoSeed administration, whichever is the longest. Male participants must not donate or bank sperm during the same time period.

      Exclusion Criteria:
* 1. Multicentric disease defined by tumours which have multiple discrete areas of contrast enhancing or non-enhancing tumour without connecting T2/ fluid-attenuated inversion recovery (FLAIR) signal abnormality. 2. Diffuse leptomeningeal disease. 3. Not eligible for surgical resection. 4. Known hypersensitivity to IRN or PLGA. 5. Prior IRN treatment (for Part 2 participants) less than 12 months from trial enrolment 6. Pregnant or lactating women or participants who intend to get pregnant during the trial.

  7. Prior active malignancy except for non-melanoma skin cancer and carcinoma in situ (of the cervix or bladder), unless diagnosed and definitively treated more than 3 years prior to surgical resection and trial drug administration. 8. Part 1 participants with relapsed GBM: treatment with another investigational drug or other intervention within 4 weeks prior to the surgical resection or 5 times the half-life (whichever is longer) before trial drug administration. 9. Part 2 participants with newly diagnosed GBM: prior RT, chemotherapy, immunotherapy, or targeted agents administered specifically for the lesion being treated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-05 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Part 1 To determine the optimal Dose of Irinotecan (RP2D) to be administered for Part 2. | 13 months
Part 2. Determination Of Progression Free Survival (PFS) to demonstrate the superiority of irinotecan-ChemoSeed compared to concurrent to SoC treatment | 39 months
  To demonstrate superiority of irinotecan-ChemoSeed concurrent to SoC treatment and administered into the resection margin following maximal safe surgical resection relative to SoC treatment alone, by assessment of progression-free survival (PFS).

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 6 months from recruitment
  ORR at 6 months by MRI using RANO 2.0 criteria, by independent central review and by investigator assessment.
Disease Control Rate (DCR) | 12 months from recruitment
  DCR at 12 months by MRI using RANO 2.0 by independent central review and investigator assessment.
Overall Survival | 39 months
  Comparison of Median OS for control and treated arms

CONTACTS AND LOCATIONS:
Overall Officials: Garth S Cruickshank, MBBS, PhD, Study Chair — Emeritus Professor of Neurosurgery, University of Birmingham UK

IPD SHARING:
Plan to Share IPD: Undecided